CLINICAL TRIAL: NCT03603184
Title: Phase III Double-blind Randomized Placebo Controlled Trial of Atezolizumab in Combination With Paclitaxel and Carboplatin in Women With Advanced/Recurrent Endometrial Cancer
Brief Title: Atezolizumab Trial in Endometrial Cancer - AtTEnd
Acronym: AtTEnd
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRFMN-EN-7556
Record Dates: First submitted 2018-05-21; First posted 2018-07-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; neoplasm; immunotherapy
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — atezolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): paclitaxel 175 mg/m2 + carboplatin AUC 5 or 6 will be administered every 21 days for 6-8 cycles or PD. Atezolizumab will be administered as I.V. infusion at a fixed dose of 1200 mg, every 21 days until objective radiological disease progression as assessed by the investigator if they do not meet any other discontinuation criteria (patient refusal, toxicity). Patients who are clinically stable at initial RECIST v 1.1 - defined progression - should continue on treatment until the next imaging assessment that should be ≥4 weeks and no longer than 8 weeks later.
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Carboplatin
- Control arm (Placebo Comparator): paclitaxel 175 mg/m2 + carboplatin AUC 5 or AUC 6 will be administered every 21 days for 6-8 cycles or PD. Placebo will be administered as I.V. infusion every 21 days until objective radiological disease progression as assessed by the investigator if they do not meet any other discontinuation criteria (patient refusal, toxicity). Patients who are clinically stable at initial RECIST v 1.1 - defined progression - should continue on treatment until the next imaging assessment that should be ≥4 weeks and no longer than 8 weeks later.
  Interventions: Drug: Placebos; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as I.V. infusion at a fixed dose of 1200 mg, every 21 days until objective radiological disease progression as assessed by the investigator if they do not meet any other discontinuation criteria (patient refusal, toxicity).
  Other Names: Tecentriq
  Arms: Experimental arm
Drug: Placebos — Placebo will be administered as I.V. infusion every 21 days until objective radiological disease progression as assessed by the investigator if they do not meet any other discontinuation criteria (patient refusal, toxicity).
  Arms: Control arm
Drug: Paclitaxel — Paclitaxel 175 mg/m2 will be administered every 21 days for 6-8 cycles or until progression of disease.
Drug: Carboplatin — Carboplatin AUC 5 or AUC 6 will be administered every 21 days for 6-8 cycles or until progression of disease.

SUMMARY:
Atezolizumab is an engineered humanised monoclonal immunoglobulin G1 antibody that binds selectively to PD-L1 and prevents its interaction with PD-1 and B7-1.

In May 2016 atezolizumab was approved by the FDA for patients with locally advanced or metastatic urothelial carcinoma who have disease progression during or following any platinum-containing chemotherapy, or within 12 months of receiving chemotherapy before surgery (neoadjuvant) or after surgery (adjuvant); in October 2016 it was approved by the FDA for patients with metastatic non-small cell lung cancer (NSCLC) who have disease progression during or following platinum-containing chemotherapy, and have progressed on an appropriate FDA-approved targeted therapy if their tumor has EGFR or ALK gene abnormalities. Finally, in April 2017 atezolizumab was granted accelerated approval by FDA for the first-line treatment of patients with locally advanced or metastatic urothelial carcinoma who are not eligible for cisplatin chemotherapy. Combinations of atezolizumab with chemotherapeutic agents and/or targeted therapies were studied in different solid tumors such as melanoma, NSCLC, renal cell carcinoma and colorectal carcinoma. From these studies the AE profile of atezolizumab combinations were consistent with that of the individual agents.

Finally, preliminary results of a Phase Ia study of Atezolizumab (NCT01375842) monotherapy in relapsed endometrial cancer were reported as abstract at ASCO 2017. Fifteen patients were evaluated for safety and efficacy with a minimum follow-up of 11.2 months. No G4-5 related AEs occurred. Regarding efficacy ORR was 13% [2/15] by RECIST. Atezolizumab seemed to have a favorable safety profile, with durable clinical benefit in some patients. Further studies with atezolizumab are warranted given its promising results in advanced endometrial cancer and the limited efficacy of current treatment options.

ELIGIBILITY:
Inclusion Criteria:

I-1. Newly diagnosed, histologically-confirmed with residual disease after surgery either measurable or evaluable, or inoperable stage III-IV endometrial carcinoma/carcinosarcoma, after diagnostic biopsy, and naïve to first line systemic anti-cancer treatment. Recurrent endometrial cancer patients if not yet treated for recurrent disease.

I-2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 I-3. Age ≥ 18 years I-4. Only one prior line of systemic platinum-based regimen is permitted if the platinum-free interval ≥ 6 months. Such prior line is the up-front/adjuvant treatment which can be concurrent chemoradiation or concurrent chemoradiation followed by chemotherapy or only chemotherapy.

I-5. Patients with history of primary breast cancer may be eligible provided they completed their definitive anticancer treatment more than 3 years ago and they remain breast cancer disease free prior to start of study treatment.

I-6. Previous pelvic and outside pelvis radiation is allowed if completed more than 6 weeks ago.

I-7. Signed informed consent and ability to comply with treatment and follow-up.

I-8. Representative FFPE tumor sample or, only if unfeasible, at least 20 unstained slides from initial surgery or from diagnostic biopsy, in case surgery was not performed, available and sent to central laboratory for Micro Satellite (MS) determination prior to randomization.

I-9. Patients must have normal organ and bone marrow function :

1. Haemoglobin ≥ 10.0 g/dL.
2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
3. Platelet count ≥ 100 x 109/L.
4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN.
6. Serum creatinine ≤ 1.5 x institutional ULN

Exclusion Criteria:

E-1. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast. Patients with a history of localized malignancy diagnosed over 5 years ago may be eligible provided they completed their adjuvant systemic therapy prior to randomization and that the patient remains free of recurrent or metastatic disease.

E-2. Patients with uterine leiomyosarcoma . E-3. Major surgery within 4 weeks of starting study treatment or patients who have not completely recovered from the effects of any major surgery.

E-4. Previous allogeneic bone marrow transplant or previous solid organ transplantation.

E-5. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted).

E-6. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD1, or anti-PDL1 therapeutic antibodies or anti-CTLA4 .

E-7. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1.

E-8. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial. However, please note that the use of inhaled corticosteroids for chronic obstructive pulmonary disease or for asthma is allowed, as well as the use of mineralocorticoids (e.g., fludrocortisones) and low-dose supplemental corticosteroids for adrenocortical insufficiency and for patients with orthostatic hypotension. The use of corticosteroids as premedication for paclitaxel-based regimen is allowed).

E-9. History of autoimmune disease, including but not limited to myasthenia gravis, myositis,autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis [please note: patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible; patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are eligible; history of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia) is permitted].

E-10. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).

E-11. Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C .

1. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive total hepatitis B core antibody [HBcAb]) are eligible only if hepatitis B virus (HBV) DNA is negative. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.
2. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.

E-12. Active tuberculosis (all patients will have tuberculin [PPD] skin test or Interferon-Gamma Releasing Assay [IGRA] done locally prior to inclusion to study) E-13. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1 E-14. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (example approximately October to March in the Northern Hemisphere). Patients must not receive live, attenuated influenza vaccine.

E-15. Clinically significant (e.g. active) cardiovascular disease, including:

1. Myocardial infarction or unstable angina within ≤ 6 months of randomization,
2. New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF),
3. Poorly controlled cardiac arrhythmia despite medication (patients with rate controlled atrial fibrillation are eligible),
4. Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision) E-16. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.

E-17. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in any case of suspected central nervous system (CNS) involvement .

E-18. History or evidence upon neurological examination of central nervous system (CNS) disease, unless asymptomatic and adequately treated with standard medical therapy.

E-19. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.

E-20. Women of childbearing potential (<2 years after last menstruation) not willing to use highly-effective means of contraception.

E-21. Pregnant or lactating women. E-22. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.

E-23. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation.

E-24. Known hypersensitivity reaction or allergy to drugs chemically related to carboplatin, paclitaxel, or their excipients that contraindicates the subject's participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
PFS in the MSI | Up to 18 months after the last patient enrolled
  PFS is defined as the time from randomization to the date of first progression or death
PFS | Up to 18 months after the last patient enrolled
  PFS is defined as the time from randomization to the date of first progression or death from any cause, whichever comes first.
  Progression will be established as the radiological disease progression according to RECIST 1.1 or death from any cause, whichever occurs first.
OS | Up to two years after the last patient enrolled
  OS is defined as the time from randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Objective response rate | Up to three years after the last patient enrolled
  Objective Response Rate (ORR), defined as the percentage of patients with an objective response as determined by RECIST 1.1
Duration of response | Up to two years after the last patient enrolled
  Duration of response, defined as the time from the date of first documentation of response (complete response (CR) or partial response (PR), whichever occurs first) to the date of documented PD or death
Safety: Maximum toxicity grade | Up to 30 days after the end of treatment
  Maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 4.03
Safety: Number of patients experiencing grade 3-4 toxicity for each toxicity | Up to 30 days after the end of treatment
  Number of patients experiencing grade 3-4 toxicity for each toxicity according to NCI-CTCAE v. 4.03
Safety: Type, frequency and nature of SAEs | Up to 30 days after the end of treatment
  Type, frequency and nature of SAEs, according to NCI-CTCAE v. 4.03
Safety: Number of patients with at least a SAE | Up to 30 days after the end of treatment
  Number of patients with at least a SAE according to NCI-CTCAE v. 4.03
Safety: Number of patients with at least a SADR | Up to two years after the last patient enrolled
  Number of patients with at least a SADR, according to NCI-CTCAE v. 4.03
Safety: Number of patients with at least a SUSAR | Up to two years after the last patient enrolled
  Number of patients with at least a SUSAR, according to NCI-CTCAE v. 4.03
Quality of life: EORTC QLQ-C30 questionnaire | Up to two years after the last patient enrolled
  Mean changes from the baseline scores in quality of life by cycle and between treatment arms.
Quality of life: QLQ-EN24 questionnaire | Up to two years after the last patient enrolled
  Mean changes from the baseline score in quality of life by cycle and between treatment arms.
Quality of life: GP5 item | Up to two years after the last patient enrolled
  Proportion of patients reporting each response option at each assessment timepoint by treatment arm for item GP5 from the FACT G instrument.
Compliance: Number of administered cycles | Up to two year after the last patient enrolled
  Number of administered cycles
Compliance: Reasons for discontinuation and treatment modification | Up to two year after the last patient enrolled
  Number of patients for each reasons
Compliance: Dose intensity | Up to two year after the last patient enrolled
  Entire dose administered during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Colombo, MD, Principal Investigator — Istituto Europeo di Oncologia (IEO) - Milan
Locations (93):
- Australia (14):
  - Royal Adelaide hospital, Adelaide
  - Border Medical Oncology Research Unit, Albury
  - Icon Cancer Centre, Auchenflower
  - Pindara Private Hospital, Benowa
  - Box Hill Hospital, Box Hill
  - Frankston Hospital, Frankston
  - Gosford Hospital, Gosford
  - Royal Brisbane and Women's Hospital, Herston
  - Royal Hobart Hospital, Hobart
  - Liverpool Hospital, Liverpool
  - Northern Cancer Institute, Saint Leonards
  - Darling Downs Hospital and Health Service - Toowoomba Hospital, Toowoomba
  - Calvary Mater Newcastle, Waratah
  - Wollongong Hospital, Wollongong
- Austria (2):
  - Medizinische Universitaet Graz - Universitätsklinik für Frauenheilkunde und Geburtshilfe, Graz
  - Medical University of Innsbruck, Innsbruck
- Germany (4):
  - Charité Universitätsmedizin Berlin, Berlin
  - Kliniken Essen Mitte, Essen
  - UniversitätsKlinikum Heidelberg, Mannheim
  - Klinikum der Ludwig-Maximilians-Universität München (LMU), München
- Italy (22):
  - AO SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Policlinico S. Orsola Malpighi, Bologna
  - Azienda Sanitaria dell'Alto Adige, Bolzano
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione Poliambulanza, Brescia
  - AOU Cagliari, Policlinico Universitario, Cagliari
  - AOU Careggi, Florence
  - ASST di Lecco, Lecco
  - Ospedale San Luca, Lucca
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Gerardo, Monza
  - Istituto Oncologico Veneto (IOV), Padua
  - AOU di Parma, Parma
  - AOU Pisana, Pisa
  - AO Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ausl Romagna, Rimini
  - Policlinico Umberto I, Università di Roma "La Sapienza", Roma
  - Ospedale di Sondrio ASST Valtellina e Alto Lario, Sondrio
  - Ospedale SS Trinità, Sora
  - AO Ordine Mauriziano, Torino
  - AOU Città della Salute e della Scienza di Torino - Ospedale Sant'Anna, Torino
  - P.O Sant'Andrea Vercelli, Vercelli
- Japan (10):
  - Hirosaki University Hospital, Aomori
  - National Cancer Center Hospital East, Chiba
  - Shikoku Cancer Center, Ehime
  - Kurume University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Tohoku University Hospital, Miyagi
  - Niigata University Medical＆Dental Hospital, Niigata
  - Osaka University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - Keio University Hospital, Tokyo
- Auckland city Hospital, Auckland, New Zealand
- South Korea (10):
  - Keimyung University Dongsan Medical Center, Daegu
  - Ilsan Cha Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (10):
  - Hospital De Sant Pau I La Santa Creu, Barcelona
  - Hospital Universitario Vall d´Hebron Institute of Oncology (VHIO), Barcelona
  - Institut Català d'Oncologia (ICO) Girona, Girona
  - Institut Català d'Oncologia (ICO), L'Hospitalet- Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Miguel Servet Zaragoza, Zaragoza
- Switzerland (8):
  - Kantonsspital, Baden
  - Universitätsspital, Basel
  - IOSI, Bellinzona
  - Inselspital, Bern
  - Kantonsspital, Lucerne
  - Frauenfeld, Münsterlingen
  - Kantonsspital, Winterthur
  - Universitätsspital, Zurich
- Taiwan (2):
  - Chang Gung Memorial Hospital-Kaohsiung, Kaohsiung City
  - Chang Gung Memorial Hospital-Linkou, Taoyuan
- United Kingdom (10):
  - Royal Derby Hospital, Derby
  - Royal Devon & Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Gartnavel General Hospital, Glasgow
  - Velindre Cancer Centre, Glasgow
  - Imperial College Healthcare NHS Trust, London
  - Royal Marsden Hospital, London
  - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - NUHT - Nottingham University Hospital NHS Trust, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harano K, Fossati R, Pardo B, Galli F, Hudson E, Antill Y, Lee C, Rabaglio M, Heitz F, Kolovetsiou-Kreiner V, Lai CH, Biagioli E, Manso L, Nishio S, Allan K, Lee YC, Uggeri S, Redondo A, Nakagawa S, Au E, Lombard J, Gadducci A, Takehara K, Baldini EE, Palaia I, Casanova C, Ardizzoia A, Bologna A, Barretina-Ginesta MP, Colombo N. Phase III double-blind randomized placebo controlled trial of atezolizumab in combination with carboplatin and paclitaxel in women with advanced/recurrent endometrial carcinoma: the Asian cohort of the AtTEnd/ENGOT-EN7 trial. J Gynecol Oncol. 2025 Jul;36(4):e117. doi: 10.3802/jgo.2025.36.e117. PMID 40590326
- [Derived] Colombo N, Biagioli E, Harano K, Galli F, Hudson E, Antill Y, Choi CH, Rabaglio M, Marme F, Marth C, Parma G, Farinas-Madrid L, Nishio S, Allan K, Lee YC, Piovano E, Pardo B, Nakagawa S, McQueen J, Zamagni C, Manso L, Takehara K, Tasca G, Ferrero A, Tognon G, Lissoni AA, Petrella M, Laudani ME, Rulli E, Uggeri S, Barretina Ginesta MP; AtTEnd study group. Atezolizumab and chemotherapy for advanced or recurrent endometrial cancer (AtTEnd): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2024 Sep;25(9):1135-1146. doi: 10.1016/S1470-2045(24)00334-6. Epub 2024 Aug 2. PMID 39102832
- [Derived] Bogani G, Monk BJ, Powell MA, Westin SN, Slomovitz B, Moore KN, Eskander RN, Raspagliesi F, Barretina-Ginesta MP, Colombo N, Mirza MR. Adding immunotherapy to first-line treatment of advanced and metastatic endometrial cancer. Ann Oncol. 2024 May;35(5):414-428. doi: 10.1016/j.annonc.2024.02.006. Epub 2024 Feb 29. PMID 38431043